CLINICAL TRIAL: NCT01494792
Title: Sofia Strep A FIA Field Study
Status: Terminated | Type: Observational
Why Stopped: Performance did not meet sponsor requirements.
Sponsor: Quidel Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-0142-02
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Group A Streptococcus; Strep Throat
MeSH Terms: interventions — Diagnosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: In Vitro Diagnositc aid for diagnosis

SUMMARY:
The purpose of this study is to demonstrate the ability of the Sofia Strep A FIA test and Sofia Analyzer to accurately detect a throat swab specimen for the presence or absence of Group A Streptococcus when compared to culture.

ELIGIBILITY:
Inclusion Criteria:

* Presence of sore throat
* Redness of the posterior pharyngeal wall
* Tonsillar exudate
* Tonsillar swelling
* Tender anterior cervical adenopathy
* Fever, > 38º C (100.4ºF) at presentation or within past 24 hours

Other symptoms that may be present, in addition to above symptoms for GAS:

* Rash, typical of scarlet fever
* Abnormal tympanic membranes
* Palatal petechiae

Exclusion Criteria:

* Subjects treated with antibiotics currently or within the previous week (7 days) are not to be included in this study.
* At clinical sites requiring informed consent, unable to understand and consent to participation; for minors this includes parent or legal guardian.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects must be three (3) years of age or older and exhibiting symptoms characteristics of pharyngitis, possibly Group A Streptococcus.
Sampling Method: Non-Probability Sample
Enrollment: 2090 (Actual)
Dates: Start 2011-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - La Costa Pediatrics, Carlsbad, California
  - Santo Nino Medical Clinic, Panorama City, California
  - La Jolla Pediatrics, San Diego, California
  - Teena Hughes, MD, Tampa, Florida
  - Children's Memorial Hospital, Chicago, Illinois
  - Twelve Corners Pediatrics, Rochester, New York
  - Montrose Family Practice, Akron, Ohio
  - Advanced Pediatrics, Vienna, Virginia